CLINICAL TRIAL: NCT00333892
Title: Leukapheresis Procedures to Obtain Lymphocytes for Research Studies on Antiretroviral Naive HIV-infected Patients
Brief Title: Leukapheresis to Obtain Lymphocytes for Studies on Antiretroviral Naive HIV-infected Patients
Status: Completed | Type: Observational
Sponsor: Canadian Immunodeficiency Research Collaborative (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 8737
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: primary HIV infection; chronic HIV infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Leukapheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Obtain lymphocytes for research studies on anti-retroviral naive HIV-infected patients.

INTERVENTIONS:
Procedure: leukapheresis — pack of cells as per protocol

SUMMARY:
To further investigate differences in the immunologic function of various lymphocyte subsets in HIV-infected patients who are treated early in their infection and during the chronic phase of the infection. Studies will also be done to further delineate the various antigen-specific and innate immune responses including characterization of soluble factors associated with primary HIV infection.

DETAILED DESCRIPTION:
Primary HIV-1 infected and chronically infected individuals will be recruited and leukapheresis will be performed. This one year study requires that patients be apheresed once before initiating therapy and on two other occasions (at month 6 and month 12) after suppression of plasma viremia. Peripheral blood mononuclear cells will be isolated by sodium diatrizoate density centrifugation and subjected to immunologic and virologic studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult HIV-1 infected patient
* For primary infected patients anyone with an exposure to a known source of HIV infected material or individual, with symptoms and signs if present consistent with primary HIV infection, a negative ELISA, indeterminate Western blot for HIV and a positive HIV plasma RNA levels > 10,000 copies/mL by either RT-PCR or bDNA
* Chronic HIV-infected patients should have a positive ELISA and a confirmatory western blot and willingness to give informed consent for the storage of blood.
* Willingness to be able to make follow-up visits for apheresis at 6 and 12 months for those who undergo antiretroviral therapy

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-infected adults who have a positive ELISA and a confirmatory western blot HIV test.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2003-08; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ostrowski, MD, Principal Investigator — University of Toronto